CLINICAL TRIAL: NCT03016273
Title: Bladder Flap Versus Non Bladder Flap Technique In Women Undergoing Elective Cesarean Section A Randomized Controlled Trial
Brief Title: Bladder Flap Technique In Elective Cesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yasmin mohamed Alaa eldin mahmoud Youssef, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BFCS
Record Dates: First submitted 2017-01-09; First posted 2017-01-10 (Estimated); Last update posted 2017-07-05 (Actual); Status verified 2017-07

CONDITIONS: Cesarean Delivery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bladder flap (Experimental): The bladder flap is made by superficially incising and dissecting the peritoneal lining to separate the urinary bladder from the lower uterine segment.
  Interventions: Procedure: creation of bladder flap
- Non bladder flap (No Intervention)

INTERVENTIONS:
Procedure: creation of bladder flap — Creation of the bladder flap, i.e., dissecting the urinary bladder from the lower segment of the uterus is a standard part of cesarean section (CS).
  Arms: Bladder flap

SUMMARY:
Cesarean section is a surgical procedure used to deliver one or more babies. cesarean section is usually performed when vaginal delivery will put the mother or child's health or life at risk. In recent years, the number of cesarean section has risen worldwide.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing elective primary cesarean section
2. previous cesarean section
3. gestational age 32 or more.

Exclusion Criteria:

1. Patients undergoing emergent cesarean section
2. Patients undergoing planned vertical uterine incision.
3. Patients undergone previous laparotomies.
4. Gestational age less than 32 weeks .
5. Patient refusing to participate in the study
6. Women with body mass index >35

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-02-20 (Actual); Primary Completion 2018-02 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
the skin - delivery time | duration of surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Assuit university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided